CLINICAL TRIAL: NCT02695212
Title: A Phase 2 Open-label Single Center Study to Evaluate the Efficacy of Apremilast for the Treatment of Moderate Hidradenitis Suppurativa
Brief Title: Single Center Study of Apremilast for the Treatment of Hidradenitis Suppurativa
Acronym: HS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Florida Academic Dermatology Centers (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AP-CL-HYDSUP-PI-004953
Record Dates: First submitted 2016-02-26; First posted 2016-03-01 (Estimated); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — apremilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Apremilast ( open label) (Experimental): Investigational Product: Apremilast
  Doses: Period A:
  10mg Per day, day #1, 10mg Twice Per day, day #2 10mg qAM, 20mg qHS day #3 20mg Twice per day, day #4 20mg qAM, 30 mg qHS day #5 30mg Twice per day, day #6
  Period B:
  30mg Twice per day, day #7 through week #24
  Period C:
  Week 28 (4 weeks off therapy), for final evaluation Mode of Administration: Oral
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: Apremilast — Investigational Product: Apremilast
  Doses: Period A:
  10mg Per day, day #1, 10mg Twice Per day, day #2 10mg qAM, 20mg qHS day #3 20mg Twice per day, day #4 20mg qAM, 30 mg qHS day #5 30mg Twice per day, day #6
  Period B:
  30mg Twice per day, day #7 through week #24
  Period C:
  Week 28 (4 weeks off therapy), for final evaluation Mode of Administration: Oral

SUMMARY:
The primary objective of this study is to evaluate the safety and efficacy of Apremilast in subjects with moderate Hidradenitis Suppurativa (HS).

DETAILED DESCRIPTION:
This study is an open-label 28-week trial. All Subjects will receive Apremilast with the initial titrating dose as per package insert (10mg per day on day #1, escalating to 30mg twice daily at day #6 and continuation at this dose).

The primary efficacy endpoint is:

The Proportion of subjects achieving Hidradenitis Suppurativa Clinical Response (HiSCR) at week 16, defined as a 30% reduction in the total number of abscess and inflammatory nodule count with a 50% reduction as an exploratory endpoint..

The Secondary endpoints are:

1. The number of patients achieving a one point reduction in the Physician's Global Assessment (PGA) score at week 16
2. Changes in Modified Sartorius scale from Baseline to Week 16
3. The number of patients achieving a two point reduction (required from baseline score) in the Visual Analog Scale (VAS) pain score at week 16
4. Dermatology Life Quality Index or DLQI,

The study will be conducted over 24 weeks on active therapy followed by a four week observational visit. The total length of the study will be 28 weeks.

Study visits will occur at Baseline (Week 0), Weeks 4, 8, 12, 16, 20, 24, and then a observational follow up 4 weeks afterwards. Additionally, all subjects will be contacted by phone 1 week following the Baseline visit to ensure daily pain assessments are being recorded. If any signs or symptoms are reported at the time of the call, an unscheduled study visit will be conducted to assess whether an infection is present.

Adverse events will be collected throughout the study.

ELIGIBILITY:
Inclusion Criteria:• Have the capacity to understand and sign and Informed Consent Form.

* Subject must be in general good health ( except for Hidradenitis Suppurativa) as judged by the Investigator, based on medical history, physical examination, clinical laboratories and urinalysis. NOTE: the definition of good health means a subjects that does not have uncontrolled significant co-morbid conditions.
* Must have a diagnosis of Hidradenitis Suppurativa (HS) for at least 6 months prior to Baseline/Screening visit
* Subjects with moderate Hidradenitis Suppurativa (HS) with a Physician's Global Assessment (PGA) score of 3 defined as having: 0 abscesses, 0 draining fistula, and 5 inflammatory nodules; or 1 abscess or draining fistula and 1 inflammatory nodule; or 2-5 abscesses or draining fistulas and 10 inflammatory nodules
* Hidradenitis Suppurativa (HS) lesions must be present in at least two distinct anatomic areas, one of which must be at least Hurley Stage II (see definition of terms)
* Subject must have stable HS for at least 2 months (60 days) prior to Screening/ Baseline visit as determined by the investigator through subject interview and review of medical history;
* Subject must have a total abscess and inflammatory nodule (AN) count (PGA) of no greater than moderate at the Baseline visit. Patient with PGA 0-1 (No disease or minimal Disease will be excluded).
* Subject must agree to daily use (and throughout the entirety of the study) of one of the following over-the-counter topical antiseptics on their Hidradenitis Suppurativa (HS) lesions: chlorhexidine gluconate, triclosan, benzoyl peroxide, or dilute bleach in bathwater.
* Women who are postmenopausal must have a negative serum pregnancy test on entry in the study.
* Females of childbearing potential (FCBP)† must have a negative pregnancy test at Screening and Baseline. While on investigational product and for at least 28 days after taking the last dose of investigational product, FCBP who engage in activity in which conception is possible must use one of the approved contraceptive§ options described below:

Option 1: Any one of the following highly effective methods: hormonal contraception (oral, injection, implant, transdermal patch, vaginal ring); intrauterine device (IUD); tubal ligation; or partner's vasectomy; OR Option 2: Male or female condom (latex condom or nonlatex condom NOT made out of natural [animal] membrane [for example, polyurethane]; PLUS one additional barrier method: (a) diaphragm with spermicide; (b) cervical cap with spermicide; or (c) contraceptive sponge with spermicide.

* Male subjects (including those who have had a vasectomy) who engage in activity in which conception is possible must use barrier contraception (male latex condom or nonlatex condom NOT made out of natural [animal] membrane [for example, polyurethane]) while on investigational product and for at least 28 days after the last dose of investigational product.

  † A female of childbearing potential is a sexually mature female who 1) has not undergone a hysterectomy (the surgical removal of the uterus) or bilateral oophorectomy (the surgical removal of both ovaries) or 2) has not been postmenopausal for at least 24 consecutive months (that is, has had menses at any time during the preceding 24 consecutive months).

  § The female subject's chosen form of contraception must be effective by the time the female subject is randomized into the study (for example, hormonal contraception should be initiated at least 28 days before randomization).
* The screening/baseline laboratory test results must meet the following criteria (WNL means within normal limits for patients with HS [e.g., may have slightly higher WBC and platelet counts]):
* WBC (white blood cell count): WNL
* ANC (absolute neutrophil count): WNL
* Hemoglobin: >10 mg/dl
* Platelets: WNL
* Serum Creatinine: WNL
* SGOT (AST - aspartate aminotransferase): <2 times upper normal limit
* SGPT (ALT - alanine aminotransferase): <2 times upper normal limit
* Alkaline phosphatase:<2 times upper normal limit

Exclusion Criteria:

* The presence of any of the following will exclude a subject from enrollment:
* Subjects with PGA 4 and 5 , with 15 lesions and significant scarring (defined as any linear, indurated area, extended across more than 50% of the circumference of the affected area) ,fistulas or sinus tract involvement will be excluded.
* Other than Hidradenitis Suppurativa , any clinically significant (as determined by the Investigator) cardiac, endocrinologic, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic disease, or other major disease that is currently uncontrolled.
* Any condition, including the presence of laboratory abnormalities, which would place the subject at unacceptable risk if he/she were to participate in the study.
* Prior history of suicide attempt at any time in the subject's life time prior to screening or randomization, or major psychiatric illness requiring hospitalization within the last 3 years.
* Women who are pregnant, nursing, or planning pregnancy within 6 months after the last study drug dose (this includes father's who plan on fathering a child within 6 months after their last study drug dose.
* Active substance abuse or a history of substance abuse within 6 months prior to Screening
* Malignancy or history of malignancy, except for:
* treated [ie, cured] basal cell or squamous cell in situ skin carcinomas;
* treated [ie, cured] cervical intraepithelial neoplasia (CIN) or carcinoma in situ of cervix with no evidence of recurrence within the previous 5 years.
* Active substance abuse or a history of substance abuse within 6 months prior to Screening. .
* Patient with diagnosis or suspected Crohns disease
* Patient who is on a stable dose of analgesics, will be allowed to remain on them. No new opiates will be permitted during the trial.
* Use of any investigational drug within 4 weeks prior to randomization, or 5 pharmocokinetic/pharmacodynamic half-lives, if known (whichever is longer).
* Prior treatment with Apremilast
* Known allergy to Apremilast
* Have a known history of serious infections (eg, hepatitis, pneumonia or pyelonephritis) in the previous 3 months
* Have a history of lymphoproliferative disease, including lymphoma or signs suggestive of possible lymphoproliferative disease such as lymphadenopathy of unusual size or location (eg, nodes in the posterior triangle of the neck, infraclavicular, epitrochlear, or periaortic area), or splenomegaly
* Have current signs or symptoms of severe, progressive or uncontrolled renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, or cerebral disease.
* Are unable or unwilling to undergo multiple venipunctures because of poor tolerability or lack of easy access
* Patient with significant scarring, fistulas, or sinus tract involvement will be excluded. Only subjects with inflammatory abscesses and nodules will be allowed to enter the study.
* Infection(s) requiring treatment with intravenous (IV) anti-infectives (antibiotics, antivirals, antifungals) within 30 days prior to Baseline or oral anti-infectives (antibiotics, antivirals, antifungals) within 14 days prior to Baseline
* Any other active skin disease or condition (e.g., bacterial, fungal or viral infection) that may interfere with assessment of HS;
* History of invasive infection (e.g., listeriosis, histoplasmosis), human immunodeficiency virus (HIV);
* Subject has an active systemic viral infection or any active viral infection that based on the investigator's clinical assessment make the subject an unsuitable candidate for the study;
* Hepatitis B: HBsAg positive (+) or detected sensitivity on the HBV-DNA PCR qualitative test for HBc Ab/HBsAb positive subjects; Or Hepatitis C
* Chronic recurring infections or active TB;
* Evidence of dysplasia
* Pregnant (or considering becoming pregnant) or lactating females.
* The use of any prior biologic therapy is prohibited
* Subjects currently undergoing any of the following treatments for HS will require a 2 week wash-out period: Minocycline; Tetracycline; Clindamycin; Rifampicin and Steroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-07; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
The Proportion of subjects achieving Hidradenitis Suppurativa Clinical Response (HiSCR) | Week 16
  defined as a 30% reduction in the total number of abscess and inflammatory nodule count with a 50% reduction as an exploratory endpoint..

SECONDARY OUTCOMES:
The number of patients achieving a one point reduction in the Physician's Global Assessment (PGA) score | Week 16
  The number of patients achieving a one point reduction in thePhysician's Global Assessment (PGA) score
Changes in Modified Sartorius scale from Baseline | From Baseline to Week 16
  Changes in Modified Sartorius scale from Baseline
3. The number of patients achieving a two point reduction (required from baseline score) in the Visual Analog Scale (VAS) pain score | Week 16
  3. The number of patients achieving a two point reduction (required from baseline score) in the Visual Analog Scale (VAS) pain score

CONTACTS AND LOCATIONS:
Locations (1):
- Florida Academic Dermatology Centers, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Statistical Analysis Plan (2018-08-06): https://cdn.clinicaltrials.gov/large-docs/12/NCT02695212/SAP_000.pdf